CLINICAL TRIAL: NCT00948402
Title: Effects of Metformin Versus Oral Contraceptives on PED/PEA-15 Protein Expression in Obese Women With Polycystic Ovary Syndrome
Brief Title: PED/PEA-15 Protein, PCOS, Obesity, Insulin Sensitivity Indexes, Metformin, Oral Contraceptives
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Annamaria Colao, Dept of Moll Clin Endocrinol Oncol, University Federico II of Naples
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NeuroendoUnit-11
Record Dates: First submitted 2009-07-24; First posted 2009-07-29 (Estimated); Last update posted 2009-10-14 (Estimated); Status verified 2009-10

CONDITIONS: Polycystic Ovarian Syndrome; Insulin Sensitivity
Keywords: PED/PEA-15 protein; PCOS; IR; metformin; OCP; Oral Contraceptive
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance | interventions — Metformin; Biguanides; Contraceptives, Oral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- metformin (Experimental)
  Interventions: Drug: Metformin
- oral contraceptive (Active Comparator)
  Interventions: Drug: oral contraceptive

INTERVENTIONS:
Drug: Metformin — metformin 1250 mg three times daily
  Other Names: Biguanides
  Arms: metformin
Drug: oral contraceptive — 30 µg ethinylestradiol plus 30 mg drospirenone 21 day/month.
  Other Names: estroprogestins
  Arms: oral contraceptive

SUMMARY:
Insulin-resistance plays an important role in polycystic ovary syndrome (PCOS) physiopathology. The phosphoprotein enriched in the diabetes (PED/PEA-15), a 15 kDa protein related to insulin sensitivity, is over-expressed in type 2 diabetic patients and in PCOS women, independently of obesity. The effectiveness of oral contraceptives pills (OCP) or metformin (MET) in PCOS management is still uncertain. Aim of this pilot clinical study was to compare the effects of OCPs or MET on the expression of PED/PEA-15 in association with insulin sensitivity in obese PCOS women. Outcome measures: PED/PEA-15, BMI, plasma glucose and insulin, 1/HOMA-IR, homeostasis model assessment of insulin resistance; QUICKI, quantitative insulin sensitivity check index; ISI: whole-body insulin sensitivity index. Study design: twenty obese PCOS women (age: 24.7±18 yr; BMI: 30±2.4 kg/m2) were randomized according to insulin sensitivity to receive 30 µg ethinylestradiol plus 30 mg drospirenone 21 day/month or MET 1250 mg three times daily for 6 months. Results: At baseline, age and BMI were not different in the two groups; PED/PEA-15 protein expression was higher in MET than in OCP group (p=0.011), along with higher 1/HOMA-IR (p=0.004), and lower QUICKI and ISI (p=0.003 and p<0.001, respectively). After treatment, independently of body weight, only in MET group PED/PEA-15 decreased (p=0.004), along with insulin and 1/HOMA-IR (p<0.001), and QUICKI and ISI increased (p<0.001). Insulin sensitivity indexes improvement correlated significantly with PED/PEA-15 protein expression, but not with BMI. Conclusions: PED/PEA-15 protein over-expression in obese PCOS women with IR reduced after a six month treatment with MET, while remained unchanged in the OCP group. The reduction was independent of body weight, and correlated with insulin sensitivity indexes. This effect further supported MET as a more effective therapy than OCPs for obese PCOS women with IR, also when fertility is not required.

DETAILED DESCRIPTION:
Subjects:

Twenty obese PCOS women (age: 24.7±18 yr; BMI: 30±2.4 kg/m2) were consecutively admitted to the Endocrinology Unit of the Department of Molecular and Clinical Endocrinology and Oncology of the Federico II University of Naples, and were enrolled in this clinical study. The diagnosis of PCOS was made according to the diagnostic criteria for PCOS At study entry the patients were randomized in two groups of treatment, according to insulin sensitivity. OCP group, 10 patients (BMI 29.7± 1.5 kg/m2) received 30 µg ethinylestradiol plus 30 mg drospirenone 21 day/month. MET group, 10 patients (BMI 30.4± 3.1 kg/m2), received metformin 1250 mg three times daily. The duration of follow-up was 6 months. The control group consisted of 10 healthy female volunteers, who were age matched.

Methods:

As all PCOS women were anovulatory, they underwent a progesterone challenge test (100 mg natural progesterone i.m.; Prontogest, Amsa, Rome, Italy), which induced uterine bleeding in all PCOS women. To exclude the presence of type 2 diabetes or abnormal glucose tolerance, the oral glucose tolerance test (OGTT) was performed and the normal glucose response to the OGTT was defined according to the 'Report of the Expert Committee on the diagnosis and classification of diabetes mellitus'.

All anthropometric measurements were taken with subjects wearing only light clothes and without shoes. In each woman, weight and height were measured to calculate the BMI [weight (kg) divided by height squared (m2), kg/m2]. Height was measured to the nearest cm using a wall-mounted stadiometer. Body weight (BW) was determined to the nearest 50 g using a calibrated balance beam scale.

Patients were given a standardized interview to obtain information about the duration of obesity, eating patterns, smok¬ing habits and physical exercise. In particular, subjects were also asked to make a daily record of the amount of physical activity (no exercise; ≤2-3 h/week; ≥2-3 h/week). Preadmission food intake and dietary history were assessed by a skilled dietitian who used a computer-assisted interview (Winfood 1.5, Medimatica srl, Martinsicuro, Italy). All PCOS women received a normo-caloric diet.

Assays:

Blood samples were obtained between 08.00 h and 09.00 h from an antecubital vein after an overnight fast, with the patient in the resting position. The OGTT was performed using 75 g dextrose. Blood samples were obtained at 0, 30, 60, 90, 120, min for plasma glucose and insulin measurements. Fasting plasma glucose (FPG) levels were determined by the glucose oxidase method immediately after the OGTT. Fasting plasma insulin (FPI) samples were promptly centrifuged, plasma was separated and stored at -20°C until assay. FPI was measured by a solid-phase chemiluminescent enzyme immunoassay using commercially available kits (Immunolite Diagnostic Products Co, Los Angeles, CA). 1/HOMA-IR, QUICKI and ISI were calculated.

PED/PEA-15 protein was measured in white-blood cells (WBC) lysates obtained from 10 to 12 ml of freshly collected uncoagulated whole blood, after separation with dextran 6%, using Western blot analysis. For Western blot analysis WBC were solubilized at 4°C in TAT buffer, centrifuged at 500g for 20 min, and supernatant fractions were stored at -20°C until used. The amount of 50 μg of lysate proteins were heated at 100°C in Laemmli buffer. Proteins were separated by 15% SDS-PAGE and then transferred to 0•45-mm Immobilon-P membranes (Millipore, Bedfort, MA). Filters were probed with PED/PEA-15 antiserum at 1:2000 dilution, revealed by enhanced chemiluminescence and autoradiography. The protein bands were quantified by laser densitometry and expressed as percentage of pixels (arbitrary units).

ELIGIBILITY:
Inclusion Criteria:

* female
* premenopausal
* obesity
* PCOS.

Exclusion Criteria:

* pregnancy
* type 2 diabetes or impaired glucose tolerance
* hypothyroidism
* hyperprolactinaemia
* Cushing's syndrome
* nonclassical congenital adrenal hyperplasia
* previous (within the last 6 months) use of oral contraceptives
* glucocorticoids
* antiandrogens
* ovulation induction agents
* antidiabetic and antiobesity drugs, or other hormonal drugs.

None of the subjects was affected by any neoplastic, metabolic, hepatic, and cardiovascular disorder or other concurrent medical illness (i.e. diabetes, renal disease, and malabsorptive disorders),acute and chronic inflammations based on medical history, physical examination, and routine laboratory tests, including measurement of oral temperature, white blood cell count and urinalysis.

Ages: 21 Years to 28 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2006-12; Primary Completion 2006-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
PED/PEA-15 protein expression | 6 months

SECONDARY OUTCOMES:
BMI, plasma glucose, plasma insulin, insulin sensitivity indexes (1/HOMA-IR, homeostasis model assessment of insulin resistance; QUICKI, quantitative insulin sensitivity check index; ISI, whole-body insulin sensitivity index). | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Annamaria Colao, MD PhD, Principal Investigator — Department of Molecular and Clinical Endocrinology and Oncology Federico II University of Naples

REFERENCES:
- [Derived] Savastano S, Di Somma C, Pizza G, De Rosa A, Nedi V, Rossi A, Orio F, Lombardi G, Colao A, Tarantino G. Liver-spleen axis, insulin-like growth factor-(IGF)-I axis and fat mass in overweight/obese females. J Transl Med. 2011 Aug 16;9:136. doi: 10.1186/1479-5876-9-136. PMID 21846339
- [Derived] Savastano S, Valentino R, Pizza G, De Rosa A, Orio F, Passaretti F, Formisano P, Lombardi G, Beguinot F, Colao A. Preliminary data on effects of metformin on PED/PEA-15 cellular levels in obese women with polycystic ovary syndrome. J Endocrinol Invest. 2010 Jul-Aug;33(7):446-50. doi: 10.1007/BF03346622. PMID 20671408